CLINICAL TRIAL: NCT03154866
Title: Ability of Lactobacillus Kefiri LKF01 (DSM32079) to Colonize the Intestinal Environment and Modify the Gut Microbiota Composition of Newborns Born by Caesarian Section
Brief Title: Lactobacillus Kefiri LKF01 (DSM32079) in Newborns Born by Caesarian Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Principal Investigator, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KEFINEO1
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Caesarean Section;Stillbirth; Microbial Colonization
Keywords: Lactobacillus kefiri LKF01 DSM32079; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus kefiri LKF01 DSM32079 (Experimental)
  Interventions: Dietary Supplement: Lactobacillus kefiri LKF01 DSM32079
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus kefiri LKF01 DSM32079 — Lactobacillus kefiri LKF01 DSM32079 in drop formulation. 5 drop/daily for 21 days
  Arms: Lactobacillus kefiri LKF01 DSM32079
Dietary Supplement: Placebo — Placebo in drop formulation. 5 drop/daily for 21 days
  Arms: Placebo

SUMMARY:
The mode of delivery affects the diversity and colonization pattern of the gut microbiota during the first year of infants' life.

Probiotics have been observed to positively influence the host's health, but to date few data about the ability of probiotics to modify the gut microbiota composition exist. 40 newborns born by elective caesarian sectional be randomized to a Lactobacillus kefiri LKF01 DSM32079 (LKEF) supplementation or placebo for 21 days. Changes in the gut microbiota composition were detected by using a Next Generation Sequencing technology.

ELIGIBILITY:
Inclusion Criteria:

* Term newborn
* Adeguate for gestational age
* Born by elective cesarean section
* Otherwise healthy newborn

Exclusion Criteria:

* major acute or chronic disease
* use of probiotics/antibiotics
* gastrointestinal malformation, cystic fibrosis, other genetic diseases
* concurrent participation in other clinical trials

Ages: 1 Hour to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Lactobacillus kefiri LKF01 DSM32079 (LKEF) in fecal sample | 21 days after supplementation start
  To evaluate the ability of Lactobacillus kefiri LKF01 DSM32079 (LKEF) to colonize the intestinal environment of newborns born by caesarian section and modify the gut microbiota composition by using a Next Generation Sequencing technology.
  Presence of Lactobacillus kefiri LKF01 DSM32079 (LKEF) in fecal sample.
Number of participants with treatment-related adverse event | During 21 days after supplementation
  A structured diary on possible treatment-related adverse event will be given to mothers.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No